CLINICAL TRIAL: NCT00617084
Title: RESOLUTE-III All-comers Trial: A Randomized Comparison of a Zotarolimus-Eluting Stent With an Everolimus-Eluting Stent for Percutaneous Coronary Intervention
Brief Title: Randomized, Two-arm, Non-inferiority Study Comparing Endeavor-Resolute Stent With Abbot Xience-V Stent
Acronym: RESOLUTE-AC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Version 1.2 - IP090
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Results first posted 2011-05-17 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Disease
Keywords: Drug Eluting Stents; Interventional Cardiology
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Resolute (Active Comparator): Medtronic Endeavor Resolute
  Interventions: Device: Medtronic Endeavor Resolute
- 2. XIENCE V (Active Comparator): Abbott Xience V
  Interventions: Device: Abbott Xience V

INTERVENTIONS:
Device: Medtronic Endeavor Resolute — Medtronic Endeavor Resolute
  Other Names: Endeavor Resolute Zotarolimus-Eluting Coronary Stent System
  Arms: 1. Resolute
Device: Abbott Xience V — Abbott Xience V
  Other Names: XIENCE V Everolimus Eluting Coronary Stent System
  Arms: 2. XIENCE V

SUMMARY:
The RESOLUTE-III Allcomers trial is a prospective, multicenter, randomized, two-arm, international, non-inferiority, open-label study with 2300 patients at 15-20 centers. The study is a "real world, all comers" study.

Primary objective: to compare the Medtronic Endeavor-Resolute (Zotarolimus-Eluting stent) system with the Abbott XIENCE V (Everolimus-Eluting stent) system with respect to cardiac death, myocardial infarction (not clearly attributable to a non-target vessel), Target Lesion Revascularization at 1 year in a "real world" patient population.

DETAILED DESCRIPTION:
The RESOLUTE-III Allcomers trial is a prospective, multicenter, randomized, two-arm, international, non-inferiority, open-label study with 2300 patients at 15-20 centers. The study is a "real world, all comers" study.

Primary objective: to compare the Medtronic Endeavor-Resolute (Zotarolimus-Eluting stent) system with the Abbott XIENCE V (Everolimus-Eluting stent) system with respect to cardiac death, myocardial infarction (not clearly attributable to a non-target vessel), Target Lesion Revascularization at 1 year in a "real world" patient population.

Study hypothesis: To determine whether the Zotarolimus-Eluting stent (Medtronic Endeavor-Resolute) is non-inferior to the Everolimus-eluting stent (Abbott XIENCE V) in terms of the primary endpoint at 12 months after stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Minimal age 18 years
* Symptomatic coronary artery disease
* Patient acceptable candidate for treatment with drug eluting stent in accordance with applicable guidelines
* Presence of one or more coronary artery stenosis >50% with reference diameter 2.25-4.0mm which can be covered by one or multiple stents
* Patient indication, lesion length and vessel diameter according to 'Instructions for Use' of study stents
* Patient is willing and able to cooperate with study procedures and required follow up visits and patient or legal representative has been informed and agrees by signing EC approved written informed consent.

Exclusion Criteria:

* Women of childbearing potential who do not have a negative pregnancy test within 7 days before procedure and women who are lactating
* Known intolerance to aspirin, clopidogrel or ticlopidin, heparin, cobalt, nickel, chromium, molybdenum, polymer coatings, Zotarolimus, Everolimus, or contrast material
* Participating in other trial before reaching primary endpoint
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy is maintained throughout the peri-surgical period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2292 (Actual)
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Serruys, MD, Principal Investigator — Erasmus MC, Thoraxcenter, Rotterdam, The Netherlands; Sigmund Silber, MD, Principal Investigator — Kardiologische Praxis und Praxisklinik, Munich, Germany; Stephan Windecker, MD, Principal Investigator — University Hospital Bern, Bern, Switzerland
Locations (1):
- Stiftung Inselspital, Department of Cardiology, Bern, Switzerland

REFERENCES:
- [Derived] Koskinas KC, Siontis GC, Piccolo R, Franzone A, Haynes A, Rat-Wirtzler J, Silber S, Serruys PW, Pilgrim T, Raber L, Heg D, Juni P, Windecker S. Impact of Diabetic Status on Outcomes After Revascularization With Drug-Eluting Stents in Relation to Coronary Artery Disease Complexity: Patient-Level Pooled Analysis of 6081 Patients. Circ Cardiovasc Interv. 2016 Feb;9(2):e003255. doi: 10.1161/CIRCINTERVENTIONS.115.003255. PMID 26823484
- [Derived] Iqbal J, Serruys PW, Silber S, Kelbaek H, Richardt G, Morel MA, Negoita M, Buszman PE, Windecker S. Comparison of zotarolimus- and everolimus-eluting coronary stents: final 5-year report of the RESOLUTE all-comers trial. Circ Cardiovasc Interv. 2015 Jun;8(6):e002230. doi: 10.1161/CIRCINTERVENTIONS.114.002230. PMID 26047993
- [Derived] Taniwaki M, Windecker S, Zaugg S, Stefanini GG, Baumgartner S, Zanchin T, Wenaweser P, Meier B, Juni P, Raber L. The association between in-stent neoatherosclerosis and native coronary artery disease progression: a long-term angiographic and optical coherence tomography cohort study. Eur Heart J. 2015 Aug 21;36(32):2167-76. doi: 10.1093/eurheartj/ehv227. Epub 2015 Jun 3. PMID 26040806
- [Derived] Campos CM, Costa F, Garcia-Garcia HM, Bourantas C, Suwannasom P, Valgimigli M, Morel MA, Windecker S, Serruys PW. Anatomic characteristics and clinical implications of angiographic coronary thrombus: insights from a patient-level pooled analysis of SYNTAX, RESOLUTE, and LEADERS Trials. Circ Cardiovasc Interv. 2015 Apr;8(4):e002279. doi: 10.1161/CIRCINTERVENTIONS.114.002279. PMID 25825008
- [Derived] Taniwaki M, Radu MD, Garcia-Garcia HM, Heg D, Kelbaek H, Holmvang L, Moschovitis A, Noble S, Pedrazzini G, Saunamaki K, Dijkstra J, Landmesser U, Wenaweser P, Meier B, Stefanini GG, Roffi M, Luscher TF, Windecker S, Raber L. Long-term safety and feasibility of three-vessel multimodality intravascular imaging in patients with ST-elevation myocardial infarction: the IBIS-4 (integrated biomarker and imaging study) substudy. Int J Cardiovasc Imaging. 2015 Jun;31(5):915-26. doi: 10.1007/s10554-015-0631-0. Epub 2015 Feb 28. PMID 25721728
- [Derived] Taniwaki M, Stefanini GG, Silber S, Richardt G, Vranckx P, Serruys PW, Buszman PE, Kelbaek H, Windecker S; RESOLUTE All-Comers Investigators. 4-year clinical outcomes and predictors of repeat revascularization in patients treated with new-generation drug-eluting stents: a report from the RESOLUTE All-Comers trial (A Randomized Comparison of a Zotarolimus-Eluting Stent With an Everolimus-Eluting Stent for Percutaneous Coronary Intervention). J Am Coll Cardiol. 2014 Apr 29;63(16):1617-25. doi: 10.1016/j.jacc.2013.12.036. Epub 2014 Feb 13. PMID 24530680
- [Derived] Silber S, Kirtane AJ, Belardi JA, Liu M, Brar S, Rothman M, Windecker S. Lack of association between dual antiplatelet therapy use and stent thrombosis between 1 and 12 months following resolute zotarolimus-eluting stent implantation. Eur Heart J. 2014 Aug 1;35(29):1949-56. doi: 10.1093/eurheartj/ehu026. Epub 2014 Feb 7. PMID 24510638
- [Derived] Richardt G, Leschke M, Abdel-Wahab M, Toelg R, El-Mawardy M, Serruys PW, Silber S, Windecker S, Belardi JA, Neumann FJ, Widimsky P; RESOLUTE All Comers; RESOLUTE International Investigators. Clinical outcomes of the Resolute zotarolimus-eluting stent in patients with in-stent restenosis: 2-year results from a pooled analysis. JACC Cardiovasc Interv. 2013 Sep;6(9):905-13. doi: 10.1016/j.jcin.2013.04.017. Epub 2013 Aug 14. PMID 23954063
- [Derived] Gutierrez-Chico JL, Raber L, Regar E, Okamura T, di Mario C, van Es GA, Windecker S, Serruys PW. Tissue coverage and neointimal hyperplasia in overlap versus nonoverlap segments of drug-eluting stents 9 to 13 months after implantation: in vivo assessment with optical coherence tomography. Am Heart J. 2013 Jul;166(1):83-94. doi: 10.1016/j.ahj.2013.04.001. Epub 2013 May 3. PMID 23816026
- [Derived] Silber S, Serruys PW, Leon MB, Meredith IT, Windecker S, Neumann FJ, Belardi J, Widimsky P, Massaro J, Novack V, Yeung AC, Saito S, Mauri L. Clinical outcome of patients with and without diabetes mellitus after percutaneous coronary intervention with the resolute zotarolimus-eluting stent: 2-year results from the prospectively pooled analysis of the international global RESOLUTE program. JACC Cardiovasc Interv. 2013 Apr;6(4):357-68. doi: 10.1016/j.jcin.2012.11.006. Epub 2013 Mar 20. PMID 23523454
- [Derived] Farooq V, Vranckx P, Mauri L, Cutlip DE, Belardi J, Silber S, Widimsky P, Leon M, Windecker S, Meredith I, Negoita M, van Leeuwen F, Neumann FJ, Yeung AC, Garcia-Garcia HM, Serruys PW. Impact of overlapping newer generation drug-eluting stents on clinical and angiographic outcomes: pooled analysis of five trials from the international Global RESOLUTE Program. Heart. 2013 May;99(9):626-33. doi: 10.1136/heartjnl-2012-303368. Epub 2013 Mar 6. PMID 23468513
- [Derived] Vranckx P, Farooq V, Garg S, Van Es GA, Silber S, Windecker S, Stone GW, Serruys PW. Different cardiac biomarkers to detect peri-procedural myocardial infarction in contemporary coronary stent trials: impact on outcome reporting. Heart. 2012 Oct;98(19):1424-30. doi: 10.1136/heartjnl-2012-302267. Epub 2012 Jul 21. PMID 22821273
- [Derived] Stefanini GG, Kalesan B, Pilgrim T, Raber L, Onuma Y, Silber S, Serruys PW, Meier B, Juni P, Windecker S. Impact of sex on clinical and angiographic outcomes among patients undergoing revascularization with drug-eluting stents. JACC Cardiovasc Interv. 2012 Mar;5(3):301-10. doi: 10.1016/j.jcin.2011.11.011. PMID 22440496
- [Derived] Gutierrez-Chico JL, Wykrzykowska J, Nuesch E, van Geuns RJ, Koch KT, Koolen JJ, di Mario C, Windecker S, van Es GA, Gobbens P, Juni P, Regar E, Serruys PW. Vascular tissue reaction to acute malapposition in human coronary arteries: sequential assessment with optical coherence tomography. Circ Cardiovasc Interv. 2012 Feb 1;5(1):20-9, S1-8. doi: 10.1161/CIRCINTERVENTIONS.111.965301. Epub 2012 Feb 7. PMID 22319063
- [Derived] Gomez-Lara J, Heo JH, Brugaletta S, Garg S, Garcia-Garcia HM, van Geuns RJ, Silber S, Windecker S, Serruys PW. Risk of target lesion failure in relationship to vessel angiographic geometry and stent conformability using the second generation of drug-eluting stents. Am Heart J. 2011 Dec;162(6):1069-1079.e2. doi: 10.1016/j.ahj.2011.09.010. Epub 2011 Nov 8. PMID 22137081
- [Derived] Gutierrez-Chico JL, Regar E, Nuesch E, Okamura T, Wykrzykowska J, di Mario C, Windecker S, van Es GA, Gobbens P, Juni P, Serruys PW. Delayed coverage in malapposed and side-branch struts with respect to well-apposed struts in drug-eluting stents: in vivo assessment with optical coherence tomography. Circulation. 2011 Aug 2;124(5):612-23. doi: 10.1161/CIRCULATIONAHA.110.014514. Epub 2011 Jul 18. PMID 21768536
- [Derived] Gutierrez-Chico JL, van Geuns RJ, Regar E, van der Giessen WJ, Kelbaek H, Saunamaki K, Escaned J, Gonzalo N, di Mario C, Borgia F, Nuesch E, Garcia-Garcia HM, Silber S, Windecker S, Serruys PW. Tissue coverage of a hydrophilic polymer-coated zotarolimus-eluting stent vs. a fluoropolymer-coated everolimus-eluting stent at 13-month follow-up: an optical coherence tomography substudy from the RESOLUTE All Comers trial. Eur Heart J. 2011 Oct;32(19):2454-63. doi: 10.1093/eurheartj/ehr182. Epub 2011 Jun 9. PMID 21659439
- [Derived] Stefanini GG, Serruys PW, Silber S, Khattab AA, van Geuns RJ, Richardt G, Buszman PE, Kelbaek H, van Boven AJ, Hofma SH, Linke A, Klauss V, Wijns W, Macaya C, Garot P, Di Mario C, Manoharan G, Kornowski R, Ischinger T, Bartorelli AL, Gobbens P, Windecker S. The impact of patient and lesion complexity on clinical and angiographic outcomes after revascularization with zotarolimus- and everolimus-eluting stents: a substudy of the RESOLUTE All Comers Trial (a randomized comparison of a zotarolimus-eluting stent with an everolimus-eluting stent for percutaneous coronary intervention). J Am Coll Cardiol. 2011 May 31;57(22):2221-32. doi: 10.1016/j.jacc.2011.01.036. PMID 21616282
- [Derived] Garg S, Serruys PW, Silber S, Wykrzykowska J, van Geuns RJ, Richardt G, Buszman PE, Kelbaek H, van Boven AJ, Hofma SH, Linke A, Klauss V, Wijns W, Macaya C, Garot P, DiMario C, Manoharan G, Kornowski R, Ischinger T, Bartorelli A, Van Remortel E, Ronden J, Windecker S. The prognostic utility of the SYNTAX score on 1-year outcomes after revascularization with zotarolimus- and everolimus-eluting stents: a substudy of the RESOLUTE All Comers Trial. JACC Cardiovasc Interv. 2011 Apr;4(4):432-41. doi: 10.1016/j.jcin.2011.01.008. PMID 21511223
- [Derived] Silber S, Windecker S, Vranckx P, Serruys PW; RESOLUTE All Comers investigators. Unrestricted randomised use of two new generation drug-eluting coronary stents: 2-year patient-related versus stent-related outcomes from the RESOLUTE All Comers trial. Lancet. 2011 Apr 9;377(9773):1241-7. doi: 10.1016/S0140-6736(11)60395-4. Epub 2011 Apr 1. PMID 21459430
- [Derived] Serruys PW, Silber S, Garg S, van Geuns RJ, Richardt G, Buszman PE, Kelbaek H, van Boven AJ, Hofma SH, Linke A, Klauss V, Wijns W, Macaya C, Garot P, DiMario C, Manoharan G, Kornowski R, Ischinger T, Bartorelli A, Ronden J, Bressers M, Gobbens P, Negoita M, van Leeuwen F, Windecker S. Comparison of zotarolimus-eluting and everolimus-eluting coronary stents. N Engl J Med. 2010 Jul 8;363(2):136-46. doi: 10.1056/NEJMoa1004130. Epub 2010 Jun 16. PMID 20554978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start recruitment: April 30, 2008 > End recruitment: October 28, 2008
  > Types of location: medical clinic
Groups:
- 1. Resolute - 12-13 Months: Medtronic Resolute - 12-13 Months
- 2. XIENCE V - 12-13 Months: Abbott Xience V - 12-13 Months
Period: Overall Study
Arm/Group | 1. Resolute - 12-13 Months | 2. XIENCE V - 12-13 Months
Started | 1140 | 1152
Completed | 1119 | 1126
Not Completed | 21 | 26
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Missed 12 Months visit | 16 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1. Resolute - 12-13 Months | 2. XIENCE V - 12-13 Months | Total
Number analyzed (Participants) | 1140 | 1152 | 2292
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 545 | 563 | 1108
  >=65 years | 595 | 589 | 1184
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (10.9) | 64.2 (10.8) | 64.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 266 | 263 | 529
  Male | 874 | 889 | 1763
Region of Enrollment [Number; unit: participants]
  Europe | 1122 | 1132 | 2254
  Middle East | 18 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Target Lesion Failure
Description: Percentage of participants that had either Cardiac Death, Myocardial Infarction (not clearly attributable to a non-target vessel)or Target Lesion Revascularization (TLR, clinically indicated) after one year. MI: Q MI if new pathological Q waves and chest pain, non Q MI if CK elevated more than two times normal, troponin elevated more than normal, according to ARC definitions. TLR, clinically indicated if associated with ischemic symptoms and angiographic min lumen diameter bigger than fifty percent by QCA or without symptoms and min lumen diameter bigger than seventy percent. Measure average.
Time Frame: 12 months
Population: Analysis per intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | 1. Resolute - 12-13 Months | 2. XIENCE V - 12-13 Months
Number analyzed (Participants) | 1140 | 1152
percentage of participants | 8.2 [8.2 to 8.2] | 8.3 [8.3 to 8.3]

2. Secondary Outcome: In-Stent Percent Diameter Stenosis
Description: In Stent Percent Diameter Stenosis at thirteen months. In Stent Percent Diameter Stenosis: measured percent of diameter stenosis at the region of the stent (calculated as 100x(RVD-MLD)/RVD using the mean values from 2 orthogonal views by QCA. RVD (Reference Vessel Diameter): average of normal segments within 10mm proximal and distal to target lesion from 2 orthogonal views using QCA. MLD (Minimal Lumen Diameter): average of 2 orthogonal views of the narrowest point wihtin the area of assessment. MLD measured during QCA by the angiographic core laboratory.
Time Frame: 13 Months
Measure: Mean (Standard Deviation); unit: Percentage diameter stenosis
Arm/Group | 1. Resolute - 12-13 Months | 2. XIENCE V - 12-13 Months
Number analyzed (Participants) | 1140 | 1152
Percentage diameter stenosis | 21.65 (14.42) | 19.76 (14.64)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | 1. Resolute - 12-13 Months | 2. XIENCE V - 12-13 Months
Serious Adverse Events (participants affected / at risk) | 435/1140 | 432/1152
Other Adverse Events (participants affected / at risk) | 0/1140 | 59/1152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Resolute - 12-13 Months (N=1140) | 2. XIENCE V - 12-13 Months (N=1152)
Anaemia (Blood and lymphatic system disorders) | 11 (15) | 7 (10)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 57 (60) | 45 (45)
Angina Pectoris (Cardiac disorders) | 89 (104) | 93 (101)
Angina Unstable (Cardiac disorders) | 27 (32) | 27 (29)
Aortic Valve Stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arteriospasm Coronary (Cardiac disorders) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 13 (18) | 16 (16)
Atrial Flutter (Cardiac disorders) | 3 (4) | 2 (2)
Atrioventricular Block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 7 (7) | 4 (4)
Bundle Branch Block Left (Cardiac disorders) | 1 (1) | 0 (0)
Bundle Branch Block Right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac Failure (Cardiac disorders) | 4 (4) | 2 (2)
Cardiac Failure Congestive (Cardiac disorders) | 7 (9) | 7 (7)
Cardiac Tamponade (Cardiac disorders) | 3 (3) | 3 (3)
Cardiogenic Shock (Cardiac disorders) | 2 (2) | 5 (5)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Congestive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cor Pulmonale Acute (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 9 (9) | 8 (9)
Coronary Artery Dissection (Cardiac disorders) | 5 (5) | 3 (3)
Coronary Artery Embolism (Cardiac disorders) | 2 (2) | 0 (0)
Coronary Artery Occlusion (Cardiac disorders) | 6 (6) | 0 (0)
Coronary Artery Perforation (Cardiac disorders) | 2 (2) | 4 (4)
Coronary Artery Restenosis (Cardiac disorders) | 2 (2) | 2 (2)
Coronary Artery Stenosis (Cardiac disorders) | 4 (4) | 3 (3)
Dressler's Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
In-Stent Coronary Artery Restenosis (Cardiac disorders) | 4 (4) | 4 (4)
Intracardiac Thrombus (Cardiac disorders) | 2 (2) | 0 (0)
Ischaemic Cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1)
Left Ventricular Failure (Cardiac disorders) | 1 (1) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 15 (16) | 9 (9)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3) | 3 (3)
Papillary Muscle Disorder (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Rub (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 3 (3)
Right Ventricular Failure (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (2) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 6 (6) | 2 (2)
Ventricular Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 5 (5)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Meniere's Disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal Disorder (Endocrine disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid Disorder (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Visual Acuity Reduced (Eye disorders) | 1 (1) | 1 (1)
Vitreous Haemorrhage (Eye disorders) | 0 (0) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 5 (5) | 6 (8)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (4)
Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 10 (10) | 16 (18)
Gastrointestinal Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (2)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatic Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chest Discomfort (General disorders) | 5 (6) | 7 (7)
Chest Pain (General disorders) | 46 (54) | 46 (50)
Death (General disorders) | 10 (10) | 14 (14)
Fatigue (General disorders) | 1 (1) | 1 (1)
Gait Disturbance (General disorders) | 1 (1) | 0 (0)
General Physical Health Deterioration (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 5 (5) | 0 (0)
Injection Site Haematoma (General disorders) | 10 (10) | 8 (11)
Injection Site Haemorrhage (General disorders) | 3 (3) | 3 (3)
Injection Site Pain (General disorders) | 1 (1) | 1 (1)
Multi-Organ Failure (General disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 2 (2) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Orthostatic Intolerance (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Unevaluable Event (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 3 (3)
Abscess Limb (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 1 (1)
Haemophilus Infection (Infections and infestations) | 0 (0) | 1 (1)
Implant Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 9 (9)
Intervertebral Discitis (Infections and infestations) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Perianal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 11 (12) | 11 (14)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 2 (2)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contrast Media Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device Malfunction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign Body Trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Implantable Defibrillator Malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple Injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pacemaker Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative Thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stent Occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombosis In Device (Injury, poisoning and procedural complications) | 8 (10) | 2 (2)
Tracheal Obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Angiogram (Investigations) | 13 (16) | 12 (18)
Arteriogram Coronary (Investigations) | 1 (1) | 1 (1)
Biopsy Lung (Investigations) | 0 (0) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1) | 1 (1)
Blood Creatine Phosphokinase MB Increased (Investigations) | 0 (0) | 4 (4)
Blood Creatinine Increased (Investigations) | 1 (1) | 1 (1)
Blood Test Abnormal (Investigations) | 1 (1) | 0 (0)
C-Reactive Protein Increased (Investigations) | 1 (1) | 0 (0)
Cardiac Enzymes Increased (Investigations) | 6 (6) | 8 (8)
Cardiac Stress Test (Investigations) | 1 (1) | 1 (1)
Cardiac Stress Test Abnormal (Investigations) | 2 (2) | 0 (0)
Carotid Pulse Decreased (Investigations) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST Segment Depression (Investigations) | 1 (1) | 2 (2)
Electrocardiogram ST Segment Elevation (Investigations) | 1 (1) | 0 (0)
Investigation (Investigations) | 1 (1) | 0 (0)
Sleep Study (Investigations) | 0 (0) | 1 (1)
Troponin I Increased (Investigations) | 3 (3) | 7 (7)
Troponin Increased (Investigations) | 0 (0) | 1 (1)
Troponin T Increased (Investigations) | 0 (0) | 2 (2)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Collagen Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (4)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign Neoplasm Of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer Female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (5)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases To Abdominal Cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urethral Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vocal Cord Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Apraxia (Nervous system disorders) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 2 (2) | 2 (2)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 3 (3) | 7 (7)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
IIIrd Nerve Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 1 (1) | 0 (0)
Partial Seizures (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Radicular Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 8 (8) | 5 (5)
Syncope Vasovagal (Nervous system disorders) | 3 (3) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 5 (5) | 3 (4)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 (0) | 2 (2)
Alcoholism (Psychiatric disorders) | 1 (4) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 4 (4)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosomatic Disease (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia, Paranoid Type (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus Urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 3 (3) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Artery Stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 9 (10) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral Stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 13 (14)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Angioplasty (Surgical and medical procedures) | 2 (2) | 0 (0)
Aortic Valve Replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Arterial Aneurysm Repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriovenous Shunt Operation (Surgical and medical procedures) | 2 (2) | 0 (0)
Baker's Cyst Excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Bladder Operation (Surgical and medical procedures) | 1 (3) | 0 (0)
Cardiac Pacemaker Insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardioversion (Surgical and medical procedures) | 0 (0) | 1 (1)
Cataract Operation (Surgical and medical procedures) | 2 (2) | 0 (0)
Colon Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary Artery Bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary Revascularisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Foot Amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hysterosalpingo-Oophorectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Ileostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Implantable Defibrillator Insertion (Surgical and medical procedures) | 4 (4) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee Meniscectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee Operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Leg Amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Meniscus Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Percutaneous Coronary Intervention (Surgical and medical procedures) | 4 (4) | 3 (3)
Preoperative Care (Surgical and medical procedures) | 0 (0) | 1 (1)
Radiotherapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Rehabilitation Therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin Graft (Surgical and medical procedures) | 1 (1) | 0 (0)
Thrombectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Toe Amputation (Surgical and medical procedures) | 0 (0) | 2 (2)
Trabeculectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 5 (6) | 0 (0)
Aortic Dissection (Vascular disorders) | 0 (0) | 1 (1)
Arterial Rupture (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 0 (0) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Essential Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Extremity Necrosis (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 2 (2)
Haemorrhage (Vascular disorders) | 7 (10) | 7 (7)
Hypertension (Vascular disorders) | 8 (8) | 4 (4)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Hypovolaemic Shock (Vascular disorders) | 0 (0) | 1 (1)
Iliac Artery Stenosis (Vascular disorders) | 0 (0) | 1 (1)
Intermittent Claudication (Vascular disorders) | 0 (0) | 1 (1)
Necrosis Ischaemic (Vascular disorders) | 1 (3) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 2 (2)
Peripheral Artery Dissection (Vascular disorders) | 2 (2) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 7 (10) | 4 (6)
Vascular Pseudoaneurysm (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Resolute - 12-13 Months (N=1140) | 2. XIENCE V - 12-13 Months (N=1152)
Chest Pain (General disorders) | 0 (0) | 59 (62)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission the Publication Committee (PC) and all co-authors will review and authorize the publication.>

* Abstracts to be submitted to the PC at least 30 days before submission for publication or presentation.>
* Manuscripts to be submitted to the PC at least 60 days before submission for publication or presentation. > The Sponsor can review results communications, and can embargo communications regarding trial results prior to public release.